CLINICAL TRIAL: NCT01062607
Title: Multinational Ambispective Study of the Clinical Management and Burden of Bipolar Disorder (WAVE bd Study)
Brief Title: Study of the Clinical Management of Bipolar Disease
Acronym: WAVE bd
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NEU-DUM-2009/1
Record Dates: First submitted 2010-01-27; First posted 2010-02-04 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Bipolar Disorders
Keywords: bipolar disorders; everyday setting; treatment adherence; global
MeSH Terms: conditions — Bipolar Disorder; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients diagnosed with Bipolar Disorder I or II (DSM-IV-TR) at any phase of the disorder with at least one mood event during the 12 months before the study start.
- 2: Patients diagnosed with Bipolar Disorder I or II (DSM-IV-TR) at any phase of the disorder with at least one mood event during the 12 months before the study start receiving Seroquel extended release at some point during the retrospective period .

SUMMARY:
This study is to provide reliable information on the management of bipolar disorders in real every day, clinical practice, to determine the clinical outcomes of such management and use of resources in relation to the disease, and to establish the factors associated with different management patterns and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Bipolar Disorder I or II (DSM-IV TR) in any phase of the disorder
* Patients who had at least one mood event (depression, mania, hypomania or mixed) according to DSM-IV TR definition during the 12 months prior to the beginning of the study

Exclusion Criteria:

* Patients who had the index mood event during the 3 months before the beginning of the study (Time 0).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bipolar patients seen in mental health centers, clinics, private settings, hospitals or specialized units
Sampling Method: Probability Sample
Enrollment: 2965 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Demographic variables | Once during study
1-year prevalence for each disease phase | everytime the patient attends the consult

SECONDARY OUTCOMES:
Use of resources | everytime the patient attends the consult
treatments prescribed, EQ5D | everytime the patient attends the consult
treatments prescribed, FAST | everytime the patient attends the consult
treatments prescribed, DAI-10 | everytime the patient attends the consult
treatments prescribed, MPR | everytime the patient attends the consult
treatments prescribed, BAS | Once during the prospective part (only if patient attends with a caregiver)

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Medina, Study Director — Medical Department.AstraZeneca Spain
Locations (213):
- Austria (5):
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Villach
  - Research Site, Vöcklabruck
  - Research Site, Wiener Neustadt
- Belgium (49):
  - Research Site, Asse
  - Research Site, Begijnendijk
  - Research Site, Berchem
  - Research Site, Bredene
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Herstal
  - Research Site, Houtvenne
  - Research Site, Ixelles-Elsene
  - Research Site, Jette
  - Research Site, Keumiée
  - Research Site, Kontich
  - Research Site, Kuringen
  - Research Site, Lebbeke
  - Research Site, Lede
  - Research Site, Lembeke
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Lubbeek
  - Research Site, Maldegem
  - Research Site, Mechelen
  - Research Site, Mol
  - Research Site, Monceau-sur-Sambre
  - Research Site, Montignies-sur-Sambre
  - Research Site, Moorsel
  - Research Site, Namur
  - Research Site, Oosteeklo
  - Research Site, Oostrozebeke
  - Research Site, Ottignies
  - Research Site, Pittem
  - Research Site, Ransart
  - Research Site, Roeselare
  - Research Site, Roux
  - Research Site, Saint-Servais
  - Research Site, Sint-Denijs-Westrem
  - Research Site, Sint-Kruis
  - Research Site, Sint-Martens-Latem
  - Research Site, Sint-Niklaas
  - Research Site, Sint-Truiden
  - Research Site, Spouwen
  - Research Site, Tienen
  - Research Site, Tournai
  - Research Site, Veurne
  - Research Site, Wezembeek-Oppem
  - Research Site, Willebroek
  - Research Site, Wilrijk
  - Research Site, Zeebrugge
  - Research Site, Zoersel
  - Research Site, Zomergem
- Brazil (13):
  - Research Site, Aparecida de Goiânia
  - Research Site, Belo Horizonte
  - Research Site, Botucatu
  - Research Site, Campinas
  - Research Site, Fortaleza
  - Research Site, Goiânia
  - Research Site, Itapira
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, São Bernardo
  - Research Site, São José
  - Research Site, São Paulo
- France (77):
  - Research Site, Ajaccio
  - Research Site, Albi
  - Research Site, Alençon
  - Research Site, Amiens
  - Research Site, Appoigny
  - Research Site, Armentières
  - Research Site, Aulnay-sous-Bois
  - Research Site, Bar-le-Duc
  - Research Site, Belfort
  - Research Site, Bergerac
  - Research Site, Besançon
  - Research Site, Blois
  - Research Site, Bordeaux
  - Research Site, Bourg-en-Bresse
  - Research Site, Bourges
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Castries
  - Research Site, Clermmont Ferrand
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Douai
  - Research Site, Esquerchin
  - Research Site, Élancourt
  - Research Site, Fains-Véel
  - Research Site, Fréjus
  - Research Site, Gap
  - Research Site, Grenoble
  - Research Site, Hauteville-Lompnes
  - Research Site, Hyères
  - Research Site, Jarnac
  - Research Site, La Charité-sur-Loire
  - Research Site, La Roche-sur-Foron
  - Research Site, La Rochelle
  - Research Site, Lavaur
  - Research Site, Le Cannet
  - Research Site, Le Havre
  - Research Site, Le Puy-en-Velay
  - Research Site, Le Vésinet
  - Research Site, Libourne
  - Research Site, Lorient
  - Research Site, Marseille
  - Research Site, Mayenne
  - Research Site, Metz
  - Research Site, Mont-de-Marsan
  - Research Site, Montberon
  - Research Site, Montpellier
  - Research Site, Montreuil
  - Research Site, Mulhouse
  - Research Site, Nancy
  - Research Site, Nanterre
  - Research Site, Nantes
  - Research Site, Neuilly-sur-Marne
  - Research Site, Nice
  - Research Site, Orsay
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Rodez
  - Research Site, Saint-Avertin
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Dizier
  - Research Site, Saint-Gratien
  - Research Site, Saint-Herblain
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Pol-sur-Ternoise
  - Research Site, Saint-Quentin
  - Research Site, Sartrouville
  - Research Site, Strasbourg
  - Research Site, Thionville
  - Research Site, Thuir
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Vendôme
  - Research Site, Versailles
  - Research Site, Wattignies
- Germany (15):
  - Research Site, Berlin
  - Research Site, Cham
  - Research Site, Dillingen
  - Research Site, Ettlingen
  - Research Site, Greifswald
  - Research Site, Grünstadt
  - Research Site, Hildesheim
  - Research Site, Karlstadt am Main
  - Research Site, Kiel
  - Research Site, Lüneburg
  - Research Site, München
  - Research Site, Regensburg
  - Research Site, Stralsund
  - Research Site, Werneck
  - Research Site, Westerstede
- Portugal (11):
  - Research Site, Angra do Heroísmo
  - Research Site, Aveiro
  - Research Site, Braga
  - Research Site, Carnaxide
  - Research Site, Coimbra
  - Research Site, Faro
  - Research Site, Lisbon
  - Research Site, Portimão
  - Research Site, Porto
  - Research Site, Setúbal
  - Research Site, Tomar
- Romania (4):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Iași
- Turkey (Türkiye) (24):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Aydin
  - Research Site, Başoğlu
  - Research Site, Bolu
  - Research Site, Bursa
  - Research Site, Çankırı
  - Research Site, D.bakir
  - Research Site, Denizli
  - Research Site, Diyarbakır
  - Research Site, Elâzığ
  - Research Site, Eskişehir
  - Research Site, Hatay
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kocaeli
  - Research Site, Manisa
  - Research Site, S.urfa
  - Research Site, Samsun
  - Research Site, Sanliurfa
  - Research Site, Sivas
  - Research Site, Tugay
  - Research Site, Yağlıca
  - Research Site, Zonguldak
- Ukraine (11):
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Luhansk
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Simferopol
  - Research Site, Vinnitsa
  - Research Site, Zaporizhzhya
- Venezuela (4):
  - Research Site, Caracas
  - Research Site, Mérida
  - Research Site, Miranda
  - Research Site, San Cristóbal

REFERENCES:
- [Derived] Vieta E, Langosch JM, Figueira ML, Souery D, Blasco-Colmenares E, Medina E, Moreno-Manzanaro M, Gonzalez MA, Bellivier F. Clinical management and burden of bipolar disorder: results from a multinational longitudinal study (WAVE-bd). Int J Neuropsychopharmacol. 2013 Sep;16(8):1719-32. doi: 10.1017/S1461145713000278. Epub 2013 May 13. PMID 23663490
- [Derived] Vieta E, Blasco-Colmenares E, Figueira ML, Langosch JM, Moreno-Manzanaro M, Medina E; WAVE-bd Study Group. Clinical management and burden of bipolar disorder: a multinational longitudinal study (WAVE-bd study). BMC Psychiatry. 2011 Apr 11;11:58. doi: 10.1186/1471-244X-11-58. PMID 21481244